CLINICAL TRIAL: NCT03233464
Title: Prevalence of Molar Incisor Hypomineralization Among a Group of Egyptian Children in Giza Governorate: A Cross Sectional Study
Brief Title: Prevalence of Molar Incisor Hypomineralization Among a Group of Egyptian Children in Giza Governorate
Acronym: MIH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Refaat Abd El-Ghaffar, Principal Investigator, Cairo University
Other Study IDs: ARefaat
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

SUMMARY:
- One single operator will assess the prevalence of molar incisor hypomineralization and its Severity among a group of Egyptian children .

DETAILED DESCRIPTION:
the study is about the prevalance of molar incisor hypomineralization and its severity among a group of Egyptian children aged 8-12 years old in Giza Governorate schools.

* Participants will be randomly selected from primary and preparatory schools in Giza governorate, seated in the school lap or an empty classroom.
* Clinical examination will be made in the daylight using disposable diagnostic sets (mirror, and explorer). No diagnostic radiographs will be taken.
* Prior to performing dental examination, index teeth including incisors and 1st permanent molars will be cleaned using a cotton roll.
* A dental explorer will be further used for cleaning molar fissures.
* The examiner carefully inspect the coronal part of the 1st permanent molars and permanent incisors for demarcated opacities.
* A specially made examination chart will be taken for the child including his name, age, address, gender, school, date, medical health and any previous dental treatment.

prevalance of molar incisor hypomineralization is measured by presence or absence.

severity is measured by Modified index based on European Academy of Paediatric Dentistry (EAPD) criteria

ELIGIBILITY:
Inclusion Criteria:

* schools in Giza Governorate.
* Positive patient acceptance for participation in the study.
* Patients who are apparently medically free from any systemic disease.

Exclusion Criteria:

* Uncooperative child.
* Children with appliances.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A group of Egyptian children aged 8-12 years old in Giza Governorate schools.
Sampling Method: Probability Sample
Enrollment: 374 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
molar incisor hypomineralization | 20 mins
  prevalance of molar incisor hypomineralization

SECONDARY OUTCOMES:
molar incisor hypomineralization | 20 mins
  severity of molar incisor hypomineralization

CONTACTS AND LOCATIONS:
Overall Officials: Aya R Abd El-Ghaffar, Bachelor, Principal Investigator — Cairo University
Locations (1):
- Aya Refaat Abd El-Ghaffar, Giza,Egypt, Egypt

REFERENCES:
- [Result] Yannam SD, Amarlal D, Rekha CV. Prevalence of molar incisor hypomineralization in school children aged 8-12 years in Chennai. J Indian Soc Pedod Prev Dent. 2016 Apr-Jun;34(2):134-8. doi: 10.4103/0970-4388.180438. PMID 27080963
- [Result] Salem K, Aziz D, Asadi M. Prevalence and Predictors of Molar Incisor Hypomineralization (MIH) among Rural Children in Northern Iran. Iran J Public Health. 2016 Nov;45(11):1528-1530. No abstract available. PMID 28032070